CLINICAL TRIAL: NCT05254223
Title: Effect of Long Term "Anti-inflammatory-diet" Advice in Patients With Rheumatoid Arthritis.
Brief Title: Anti-Inflammatory Diet Effect in Rheumatoid Arthritis Patients
Acronym: AIDE-RAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jose manuel Lou Bonafonte (Other)
Collaborators: Universidad de Zaragoza (Other); Centro de Investigación Biomédica en Red de la Obesidad y Nutrición. ISCIII (Unknown); Instituto Agroalimentario de Aragón (IA2). (Unknown); Hospital San Jorge (Huesca) (Unknown)
Responsible Party: Sponsor-Investigator, Jose manuel Lou Bonafonte, Principal Investigator, Instituto de Investigación Sanitaria Aragón
Organization: Instituto de Investigación Sanitaria Aragón (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NSP-2016-1
Record Dates: First submitted 2022-01-13; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Diet; Antiinflammatory diet; Nutrition
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Diet (NDA) (Experimental): No dietary advice (NDA)
  Interventions: Other: Control Diet
- Anti-inflammatory Diet (AIDA) (Experimental): Anti-inflammatory Dietary advice (AIDA)
  Interventions: Other: Antiinflammatory Diet

INTERVENTIONS:
Other: Antiinflammatory Diet — The intervention group is recommended to follow a diet, inspired in mediterranean diet, rich in anti-inflammatory foods. They are provided with a table with the recommended foods as well as the frequency of daily/weekly/biweekly consumption.
  Arms: Anti-inflammatory Diet (AIDA)
Other: Control Diet — The control group is recommended to follow their usual diet. Only in the case of detecting a serious nutritional problem the participant is recommended to correct it with the appropriate advice of the nutritionist.
  Arms: Control Diet (NDA)

SUMMARY:
The current study pretends to clarify, whether or not a healthy anti inflammatory diet improves different health-related outcomes in participants with rheumatoid arthritis.

DETAILED DESCRIPTION:
The current study pretends to clarify, whether or not a healthy anti-inflammatory diet improves different health-related outcomes: clinical, analytical, anthropometric and psychological outcomes in participants with rheumatoid arthritis. Due to the intervention has been based in a dietary advise, one of the goals of this study is also to evaluate the role of dietary advice in changing effectively the dietary patterns of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patients

Exclusion Criteria:

Any additional pathology or situation that could be considered, according to clinical criteria, of risk for the patient or for the study. for example:

* Chronic renal failure
* Liver failure
* Heart failure
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Changes in disease activity | Day 0, month 4, month 8 and month12.
  Disease activity is determined by Simplified Disease Activity Index (SDAI)
Changes in disease activity | Day 0, month 4, month 8 and month12.
  Disease activity is determined by DAS28 score_ c reactive protein (DAS28-CRP)
Changes in disease activity | Day 0, month 4, month 8 and month12.
  Disease activity is determined by DAS28 score_ erythrocyte sedimentation rate (DAS28-ESR)
Changes in disease activity | Day 0, month 4, month 8 and month12.
  Disease activity is determined by Clinical Disease Activity Index (CDAI)
Changes in functional capacity | Day 0, month 4, month 8 and month12.
  Functional capacity is assessed by the Health Assessment Questionnaire (HAQ).
Changes in self-perceived health | Day 0, month 4, month 8 and month12.
  Self-perceived health is evaluated by questionnaire EuroQol-5D-3L (EQ-5D)
Global analysis of the dietary pattern during the intervention (FFQ) | Month 12.
  Global analysis of the dietary pattern during the intervention is evaluated by the food frequency questionaire (FFQ)
Detailed analysis of diet. | Day 0, month 4, month 8 and month12.
  Detailled analysis of diet is carried out by 24 hour dietary recall 3 days/week. Diet will be analyzed by HD-ENRICA diet analisys software (v17). Data analyzed will be: Energy (Kcal), Proteins (g), Carbohydrates (g), Fats (g), Fibre (g), vitamins (mg), minerals (mg), water (ml).
Changes in Mediterranean Diet Adherence Score (MEDAS) | Day 0, month 4, month 8 and month12.
  Changes in MEDAS are carried out by MEDAS. 0 points means no adherence, 14 points means maximal adherence.
Changes in Dietary inflammatory Index (DII) | Day 0, month 4, month 8 and month12.
  Dietary inflammatory index are calculated with the information provides by 24 hour dietary recall 3 days/week.

SECONDARY OUTCOMES:
Changes in self-reported pain, | Every week from day 0 and during 12 months.
  Participants report weekly self perception about pain, answering to a visual analogical scale where 0 means no pain and 10 is the maximum pain imaginable.
Changes in self-reported stiffness. | Every week from day 0 and during 12 months.
  Participants report weekly self perception about stiffness answering to a scale where 0 means no stiffness and 10 is the maximum stiffness imaginable.
Changes in self-reported inflammation | Every week from day 0 and during 12 months.
  Participants report weekly self perception about inflammation answering to a scale where 0 means no stiffness and 10 is the maximum stiffness imaginable.
Changes in Lipidomics profile | Day 0, month 4, month 8 and month12.
  Lipidomics profiling will be determined by plasma gas chromatography mass spectrometry (GC/MS). Lipidomics profiling in serum samples will be correlated with lipid intake.
Changes in cytokines/Interleukins (ILs) | Day 0, month 4, month 8 and month12.
  IL-1B, IL-4, IL-6, IL-10, IL-17, TNF-a, MCP1 will be analyzed by multiplex assay. Results will be correlated with Disease activity Indexes/scores.
Changes in anthropometric mesurements | Day 0, month 4, month 8 and month12.
  Participant's height (m) and weight (Kg) will be measured and body mass index (BMI) will be calculated.
Changes in anthropometric measurements | Day 0, month 4, month 8 and month12.
  Body fat percentage (BFP) analyzed by bioelectrical impedance analysis (BIA).
Changes in anthropometric measurements | Day 0, month 4, month 8 and month12.
  Body fat percentage (BFP) analyzed by anthropometric analysis acording to ISAK procedures (international standards for anthropometric assessment ) and using Siri formula where Fat %= [(4,95/density) - 4,5] * 100

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ISAK. (2011). International Standards For Anthropometric Assessment. International Society for the Advancement of Kinanthropometry.
- [Background] Siri WE. Body composition from fluid spaces and density: analysis of methods. 1961. Nutrition. 1993 Sep-Oct;9(5):480-91; discussion 480, 492. No abstract available. PMID 8286893
- [Background] Aletaha D, Landewe R, Karonitsch T, Bathon J, Boers M, Bombardier C, Bombardieri S, Choi H, Combe B, Dougados M, Emery P, Gomez-Reino J, Keystone E, Koch G, Kvien TK, Martin-Mola E, Matucci-Cerinic M, Michaud K, O'Dell J, Paulus H, Pincus T, Richards P, Simon L, Siegel J, Smolen JS, Sokka T, Strand V, Tugwell P, van der Heijde D, van Riel P, Vlad S, van Vollenhoven R, Ward M, Weinblatt M, Wells G, White B, Wolfe F, Zhang B, Zink A, Felson D. Reporting disease activity in clinical trials of patients with rheumatoid arthritis: EULAR/ACR collaborative recommendations. Ann Rheum Dis. 2008 Oct;67(10):1360-4. doi: 10.1136/ard.2008.091454. PMID 18791055
- See also: ResearchGate is a European commercial social networking site for scientists and researchers to share papers, ask and answer questions, and find collaborators. — http://www.researchgate.net/project/Study-of-the-diet-in-rheumatoid-arthritis-patients-Evaluation-of-a-proposed-anti-inflammatory-diet